CLINICAL TRIAL: NCT06546839
Title: Comparison of Serratus Posterior Superior Interfacial Plane Block vs Serratus Anterior Plane Block on Postoperative Analgesia in Patients Underwent Video-Assisted Thoracoscopic Surgery: A Randomized, Prospective, Controlled Study
Brief Title: SPSIPB vs SAPB for Thoracoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Bahadir Ciftci, Principal Investigator, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Medipol Hospital 38
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Lung Diseases; Lung Cancer; Lung Neoplasms; Lung Cancer Metastatic; Thoracic Diseases; Thoracic Cancer; Thoracic Neoplasms
Keywords: Video assisted thoracic surgery; Postoperative analgesia management; Serratus anterior plane block; Serratus Posterior Superior Interfascial Plane Block
MeSH Terms: conditions — Lung Diseases; Lung Neoplasms; Thoracic Diseases; Thoracic Neoplasms

STUDY DESIGN:
Intervention Model Description: There are two models for this study. The first group is the SPSIPB group. The second one is the SAPB group.
Who Masked: Participant, Outcomes Assessor
Masking Description: The anesthesiologist who performs postoperative pain evaluation and the patient will not know the group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group SPSIPB = SPSIPB group (Active Comparator): SPSIPB will be performed
  Interventions: Drug: SPSIPB blcok; Drug: Postoperative analgesia management
- Group SAPB = SAPB group (Active Comparator): SAPB will be performed
  Interventions: Drug: SAPB block; Drug: Postoperative analgesia management

INTERVENTIONS:
Drug: SPSIPB blcok — A high-frequency linear US probe (11-12 MHz, Vivid Q) will be covered with a sterile sheath, and an 80 mm block needle (Braun 360°) will be used. The procedure will be performed with the patient in the lateral decubitus position. After the scapula is shifted slightly laterally, the US probe is placed sagittal at the upper corner of the spina scapula, and the serratus posterior superior muscle is visualized with the third rib. The in-plane technique will be used. The block needle will be advanced in the craniocaudal direction to enter between the serratus posterior superior and the third rib. The block location will be confirmed by injecting 5 ml of saline between the rib and the muscle. After the block location is confirmed, 30 ml of 0.25% concentration bupivacaine will be used.
  Arms: Group SPSIPB = SPSIPB group
Drug: SAPB block — In the lateral decubitus position, US probe will be placed in a sagittal plane over the midclavicular region of the thoracic cage. Then the 7th rib will be identified in the midaxillary line, followed by the identification of the following muscles overlying the 6th rib: the latissimus dorsi (superficial and posterior), teres major (superior), and serratus muscle (deep and inferior). The needle will be inserted in-plane concerning the ultrasound probe targeting the plane superficial to the serratus anterior muscle. 5 ml saline will be injected for correction. Following confirmation of the correct position of the needle, 30 ml %0.25 bupivacaine will be administered for the block.
  Arms: Group SAPB = SAPB group
Drug: Postoperative analgesia management — Patients will be administered ibuprofen 400 mgr IV every 8 hours in the postoperative period. A patient-controlled device prepared with 10 mcg/ ml fentanyl will be attached to all patients with a protocol including 10 mcg bolus without infusion dose, 10 min lockout time, and 4-hour limit. If the NRS score is ≥ 4, 0.5 mg kg-1 iv meperidine will be administered as a rescue analgesic. Postoperative patient evaluation will be performed by an anesthesiologist blinded to the procedure.

SUMMARY:
Video-assisted thoracic surgery (VATS) has recently been evaluated as the standard surgical procedure for lung surgery. Although VATS is less painful than thoracotomy, patients may feel severe pain during the first hours of the postoperative period. Analgesia management is very important for these patients in the postoperative period since insufficient analgesia can cause pulmonary complications such as atelectasis, pneumonia, and increased oxygen consumption. Ultrasound (US) guided serratus posterior superior block (SPSPB) is a new interfacial plane block defined by Tulgar et al in 2023. It is based on injection on the serratus posterior superior muscle at the level of the 2nd or 3rd rib. This block provides analgesia in conditions such as interscapular pain, chronic myofascial pain syndromes, scapulocostal syndrome, and shoulder pain. The SPS muscle is located at the C7-T2 level. It attaches to the lateral edges of the second and fifth ribs. It is innervated by the lower cervical and upper intercostal nerves. With the SPS block, these nerves are blocked and analgesia is provided. It has been reported that SPSIPB provides effective analgesia after VATS. US-guided serratus anterior plane (SAP) block provides effective analgesia in the thorax's anterior, posterior, and lateral dermatomes. It has been reported that SAP block provides effective postoperative pain management following thoracotomy, breast surgery and VATS. There is no clinical randomized study in the literature evaluating the efficacy of SPSIPB and SAP block following VATS.

DETAILED DESCRIPTION:
Video-assisted thoracic surgery (VATS) has started to be considered the standard surgical procedure for lung surgery in recent years. The advantages of VATS compared to open thoracotomy are rapid recovery, shorter hospital stays, and low risk of complications. Although it is a less painful surgical procedure compared to thoracotomy, severe acute postoperative pain can be observed especially in the first hours after VATS. Thoracic epidural analgesia (TEA), which is the gold standard for post-thoracotomy analgesia, is used in analgesia after VATS. However, due to the difference in surgical technique and trauma between open surgery and VATS, what should be the gold standard for analgesia after VATS is a matter of debate. It is supported that less invasive analgesic techniques should be applied for minimally invasive surgical procedures, especially due to the difficulty of applying TEA and its side-effect profile. Thoracic paravertebral block (TPVB) is considered the first-line regional technique for VATS surgery. However, it is difficult to apply due to its anatomical proximity to important structures such as the pleura and central neuraxial system, and it may cause complications such as pneumothorax and vascular injury. Analgesia management is very important in these patients, as insufficient analgesia in the postoperative period may cause pulmonary complications such as atelectasis, pneumonia, and increased oxygen consumption.

Ultrasound (US) guided serratus posterior superior block (SPSPB) is a new interfacial plane block defined by Tulgar et al in 2023. It is based on injection on the serratus posterior superior muscle at the level of the 2nd or 3rd rib. This block provides analgesia in conditions such as interscapular pain, chronic myofascial pain syndromes, scapulocostal syndrome, and shoulder pain. The SPS muscle is located at the C7-T2 level. It attaches to the lateral edges of the second and fifth ribs. It is innervated by the lower cervical and upper intercostal nerves. With the SPS block, these nerves are blocked and analgesia is provided.

In the cadaveric study of Tulgar et al., it was determined that the spread of serratus posterior superior interfacial plane block; 7-10 intercostal levels on the left side only in the superficial fascia of the trapezius muscle. Spread dye was observed at intercostal levels, absent on the right. There was prominent staining on both sides of the deep trapezius muscle. Both the surface and skin of the rhomboid major were stained, while the rhomboid minor was only stained in the skin. SPSP block will provide successful analgesia in procedures involving the thoracic region such as chronic myofascial pain, breast surgery, thoracic surgery, and shoulder surgery. There is no randomized study in the literature evaluating the effectiveness of SPSP block for postoperative analgesia management after VATS.

US-guided serratus anterior plane (SAP) block is an interfascial plane block and was described by Blanco in 2013. A local anesthetic solution is performed into the fascial plane of the serratus anterior muscle. It is easy to perform and has low complication rate because it is far away from the important neurological and vascular structures. The serratus anterior muscle may be seen easily with US guidance in the mid-axillary line. It provides effective analgesia in anterior, posterior, and lateral dermatomes of the thorax. It has been reported that SAP block provides effective postoperative pain management following thoracotomy, breast surgery, and VATS. There is no clinical randomized study in the literature evaluating the efficacy of SPSIPB and SAP block following VATS.

This study aims to compare US-guided SPSIPB and SAP block for postoperative analgesia management after VATS. The primary aim is to compare postoperative opioid consumption and the secondary aims are to evaluate postoperative pain scores (NRS), adverse effects related with opioids (allergic reaction, nausea, vomiting) and complications due to blocks (pneumothorax, hematoma).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) classification I-III
* Scheduled for VATS under general anesthesia

Exclusion Criteria:

history of bleeding diathesis, receiving anticoagulant treatment, known local anesthetics and opioid allergy, infection of the skin at the site of the needle puncture, pregnancy or lactation, patients who do not accept the procedure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-08-10 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
Opioid consumption (Fentanyl PCA) | Changes from baseline opioid consumption at postoperative 1, 2, 4, 8, 16 and 24 hours.
  The primary aim is to compare postoperative opioid consumption from the PCA device.

SECONDARY OUTCOMES:
Pain scores (Numerical rating scale-NRS) | Changes from baseline pain scores at postoperative 1, 2, 4, 8, 16 and 24 hours
  The secondary aim is to compare NRS at the postoperative 24 h. Postoperative pain assessment will be performed using the NRS (0 = no pain, 10 = the most severe pain felt). The NRS scores will be recorded
Need for rescue analgesia (meperidine) | Postoperative 24 hours period
  The secondary aim is to compare rescue analgesia used in the postoperative 24 h.
Adverse events | Postoperative 24 hours period
  The secondary aim is to compare the adverse events (nausea, vomiting, itching) related to opioid use

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We will not plan to share IPD

REFERENCES:
- [Background] Tulgar S, Ciftci B, Ahiskalioglu A, Bilal B, Sakul BU, Korkmaz AO, Bozkurt NN, De Cassai A, Torres AJ, Elsharkawy H, Alici HA. Serratus Posterior Superior Intercostal Plane Block: A Technical Report on the Description of a Novel Periparavertebral Block for Thoracic Pain. Cureus. 2023 Feb 3;15(2):e34582. doi: 10.7759/cureus.34582. eCollection 2023 Feb. PMID 36883093
- [Background] Ciftci B, Alver S, Ahiskalioglu A, Bilal B, Tulgar S. Serratus posterior superior intercostal plane block for breast surgery: a report of three cases, novel block and new indication. Minerva Anestesiol. 2023 Nov;89(11):1054-1056. doi: 10.23736/S0375-9393.23.17432-3. Epub 2023 Jun 1. No abstract available. PMID 37272274
- [Background] Ciftci B, Alver S, Ahiskalioglu A, Bilal B, Tulgar S. Serratus posterior superior intercostal plane block: novel thoracic paraspinal block for thoracoscopic and shoulder surgery. Minerva Anestesiol. 2024 Apr;90(4):345-347. doi: 10.23736/S0375-9393.23.17827-8. Epub 2024 Jan 19. No abstract available. PMID 38240640
- [Background] Avci O, Gundogdu O, Balci F, Tekcan MN, Ozbey M. Efficacy of serratus posterior superior intercostal plane block (SPSIPB) on post-operative pain and total analgesic consumption in patients undergoing video-assisted thoracoscopic surgery (VATS): A double-blinded randomised controlled trial. Indian J Anaesth. 2023 Dec;67(12):1116-1122. doi: 10.4103/ija.ija_589_23. Epub 2023 Dec 13. PMID 38343684